CLINICAL TRIAL: NCT05318586
Title: Effect of Individualized rTMS Based on fNIRS on the Upper Limb Spasticity After Stroke
Brief Title: Individualized rTMS Based on fNIRS to Spasticity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022JQ-982
Record Dates: First submitted 2022-03-29; First posted 2022-04-08 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-03

CONDITIONS: Stroke; Spasticity, Muscle; Rehabilitation
Keywords: Stroke; Spasticity, Muscle; Rehabilitation; fNIRS; rTMS; Activation; Brain network
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized rTMS based on fNIRS (Experimental): Low-frequency rTMS will be given to the most active brain regions assessed by fNIRS.
  Interventions: Procedure: individual rTMS based on fNIRS
- Traditional rTMS strategy (Active Comparator): The control group will always be given low-frequency rTMS to contralesional M1
  Interventions: Procedure: Traditional rTMS strategy

INTERVENTIONS:
Procedure: individual rTMS based on fNIRS — The rTMS parameters will be set according to fNIRS results.
  Arms: Individualized rTMS based on fNIRS
Procedure: Traditional rTMS strategy — The low-frequency rTMS to contralesional M1 will always be used.
  Arms: Traditional rTMS strategy

SUMMARY:
Stroke is of high morbidity and mortality, and surviving patients are often unable to take care of themselves because of severe motor dysfunction. The brain has plasticity, and makes adaptive changes after stroke, resulting in the reorganization and compensation of neural networks. However, the muscle tone of some patients will significantly increase during the recovery process, which affects the rehabilitation effect. Neuromodulation techniques such as repetitive transcranial magnetic stimulation (rTMS) have been widely used to promote brain network remodeling after stroke. The investigators attempted to evaluate the motor brain network characteristics of spastic patients by fNIRS, and used the most active brain regions as rTMS stimulation regions to evaluate the improvement effect of this individualized treatment on post-stroke spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-79 years;
* Patients with first-onset stroke within 1 to 3 months after onset;
* Consciousness, sitting balance level 1 or above, can cooperate with fNIRS assessment;
* The patient or its authorized agent signs the informed consent form.

Exclusion Criteria:

* Previous seizures;
* Suffered from mental illness such as depression, anxiety, mania, and schizophrenia before the stroke onset;
* Patients with metal on the head, cochlear implants, intracranial infections, etc. who are not suitable for rTMS.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-04-10 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
modified Ashworth scale | 1 month
  The range is 0-Ⅳ level, the higher the level, the higher the spasticity.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment of upper limb motor function | 1 month
  The score range is 0-66 points, the higher the score, the better the motor function of upper limb.
Barthel index | 1 month
  The score range is 0-100 points, the higher the score, the better the activities of daily living.
average weighted clustering coefficient | 1 month
  This is a brain network indicator based on graph theory. It is a measure of the local separation of the graph. The higher the average weighted clustering coefficient, the higher the degree of segregation of the brain network.
global efficiency | 1 month
  This is a brain network indicator based on graph theory. It is a measure of the local integration of the graph. The higher the global efficiency, the stronger the ability of the network to transmit information.
inter-density | 1 month
  It is a brain network indicator based on graph theory and is defined as the ratio of the actual number of connections among all possible connections between bilateral hemispheres.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China